CLINICAL TRIAL: NCT06143579
Title: FOLFOX-Hepatic Arterial Infusion Chemotherapy (HAIC) Combined With Lenvatinib and Envolizumab in Potentially Resectable Hepatocellular Carcinoma:A Single-arm, Open-label, Single Center, Phase II Trial
Brief Title: A Study of HAIC Combined With Lenvatinib and Envolizumab in Potentially Resectable Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhongguo Zhou, Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2023-561-01
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Potentially Resectable Hepatocellular Carcinoma
Keywords: HAIC; Lenvatinib; Envolizumab; PD-L1; TKI; potentially resectable HCC
MeSH Terms: interventions — envafolimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): FOLFOX-HAIC + Lenvatinib + Envolizumab
  Interventions: Drug: FOLFOX-HAIC+Lenvatinib+Envolizumab

INTERVENTIONS:
Drug: FOLFOX-HAIC+Lenvatinib+Envolizumab — FOLFOX-HAIC: Oxaliplatin 130 or 85 mg/m2; leucovorin 200 mg/m2; fluorouracil 400 mg/m2 intravenous bolus followed by fluorouracil 2400 mg/m2 continuous infusion over 23 hours, Q3W, 2 to 4 cycles;
  Lenvatinib: 8 mg/day (BW < 60 kg) or 12 mg/day (BW ≥ 60 kg), PO, 3-4 cycles;
  Envolizumab: 300 mg, SC, Q3W, 3-4 cycles.
  Other Names: KN035

SUMMARY:
This is a single term, open label, single Center, Phase II Trial. The study is to explore the efficacy and safety of FOLFOX-HAIC combined with Lenvatinib and Envolizumab in the treatment of patients with potentially resectable HCC.

DETAILED DESCRIPTION:
At present, surgery is the preferred modality for the treatment of HCC patients with radical cure and long-term survival. However, 70% to 80% of HCC is advanced, and only 15% to 30% of patients are able to undergo surgical resection. For unresectable HCC, transformation therapy is currently used, and the response rate can be effectively increased through the "TKI plus IO" or "TKI plus IO and local therapy" regimen. For locally advanced HCC (stage III-IV), HAIC or HAIC + systemic therapy is recommended. And the first-line treatment of advanced HCC, TKI (Lenvatinib, Donafenib) or IO combined TKI are recommended. For patients with potentially resectable HCC, there are currently few explorations, and more effective treatment options and evidence-based medical evidence are needed. Therefore, this study investigated the efficacy and safety of FOLFOX-HAIC combined with Lenvatinib and Envolizumab in the treatment of patients with potentially resectable HCC, and explored the relationship between biomarkers, prognostic factors and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have signed ICF and are able to perform follow-up visits and relevant procedures required in the protocol;
2. Age ≥ 18 years (at the time of signing the ICF);
3. Clinically, histologically or pathologically confirmed hepatocellular carcinoma without extrahepatic metastases;
4. No previous treatment containing PD- (L) 1 inhibitor and Lenvatinib;
5. Potentially resectable HCC: (1)At least one measurable lesion (according to RECIST 1.1 criteria); (2)Patients with stage IIb/IIIa (equivalent to BCLC B/C) with portal vein tumor thrombus (according to Japanese PVTT grading criteria Vp3-Vp4) or more than three tumor nodules; (3)According to the assessment of the site multidisciplinary team (MDT), like surgical resection is not currently the treatment of choice;
6. ECOG score: 0 ~ 1;
7. Child-Pugh score of ≤ 7
8. Estimated survival of more than 6 months;
9. Vital organ function meets the following requirements: (1) Blood routine: Absolute neutrophil count (ANC) ≥ 1.5 × 109/L; Platelet count (PLT) ≥ 100 × 109/L; Hemoglobin (HGB) ≥ 90 g/L; (2) Liver function: Serum creatinine (Cr) ≤ 1.5 × upper limit of normal (ULN) or clearance of creatinine ≥ 50 mL/min (Cockcroft-Gault formula); Total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN); Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) levels ≤ 2.5 × upper limit of normal (ULN); (3) Kidney function: Urine protein < 2 +; if urine protein ≥ 2 +, 24-h urine protein quantitation test result should be ≤ 1 g;
10. Normal coagulation function, no active bleeding and thrombosis (1) International normalized ratio (INR) ≤ 1.5 × ULN; (2) Active partial thromboplastin time (APTT) ≤ 1.5 × ULN; (3) Prothrombin time (PT) ≤ 1.5 × ULN;
11. Female patients of childbearing age or male patients with female sexual partners of childbearing age should take effective contraceptive measures during study treatment and for 3 months after the end of study treatment; serum or urine HCG tests must be negative and must be non-lactating within 7 days before study enrollment;
12. Patients should be compliant and cooperative with safety and survival follow-up.

Exclusion Criteria:

1. Participate in other interventional clinical studies;
2. Previous or concurrent other malignancies;
3. History of liver transplantation or undergo liver transplantation;
4. History of hypersensitivity to macromolecular protein preparations, the study drug or any of the excipients;
5. Active autoimmune disease or history of autoimmune diseases (such as the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism, previous thyroid surgery); Require bronchodilators for medical intervention of asthma; the patient has vitiligo or has complete remission of asthma in childhood, no intervention is required after adults can be included;
6. Use immunosuppressive agents, or systemic or absorbable local hormone therapy to achieve immunosuppressive purposes (dose > 10 mg/day prednisone or other effective hormones), and continue to use within 2 weeks before enrollment;
7. Uncontrolled cardiac clinical symptoms or diseases, for example: (1) NYHA class 2 or higher heart failure;(2) Unstable angina pectoris; (3) Myocardial infarction within 1 year; (4) Clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention;
8. Use traditional Chinese medicine immunomodulator within 2 weeks before enrollment;
9. Severe active infection or unexplained fever > 38.5 degrees during screening and before the first dose (subjects can be enrolled due to tumor-induced fever at the investigator discretion);
10. Congenital or acquired immunodeficiency: (1)HIV infection; (2)Active hepatitis (hepatitis B reference: HBV DNA ≥ 1000 IU/mL; hepatitis C reference: HCV RNA ≥ 1000 IU/mL); chronic hepatitis B virus carriers, HBV DNA < 2000 IU/ml, must receive concurrent antiviral therapy during the trial to be enrolled;
11. Live vaccines less than 4 weeks prior to study medication or likely during the study;
12. History of psychiatric drug abuse, alcoholism, or drug abuse;
13. Chinese herbal medicine within 4 weeks prior to first treatment;
14. Factors that may cause forced halfway termination of this study, such as other serious diseases (including mental illness) requiring concomitant treatment, serious laboratory abnormalities, accompanied by family or social factors, which may affect the subject' s safety, the collection of data and samples, or other circumstances which are unsuitable for subject enrollment as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-12-15 (Estimated); Primary Completion 2025-03-03 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
AEs | Up to 60 days after last treatment or 30 days after surgery
  Defined as the proportion of patients with AE, treatment-related AE (TRAE), immune-related AE (irAE), serious adverse event (SAE), assessed by NCI CTCAE v5.0
Overall response rate (ORR) | At the end of Cycle 4 (each cycle is 21 days)
  Defined as proportion of patients who have a best response of CR or PR

SECONDARY OUTCOMES:
Pathological complete response (pCR) | At the end of the surgery
  According to post-operative pathology, the proportion of tumor necrosis, viable. tumor cells, and tumor infiltrating lymphocytes indicated by surgical resected specimens.
Major Pathological Response(MPR) | At the end of the surgery
  Survival tumor ≤10% after surgery
R0 resection rate | At the end of the surgery
  The tumor was completely removed during surgery, and the resection margin was negative when observed microscopically without residual components of the tumor
1-year recurrence-free survival(RFS) rate | Up to one years
  Subjects underwent radical resection from the start until the date of the first documented tumor into recurrence or death from any cause in, whichever occurred first within 1 year after surgery
Recurrence-free survival(RFS) | Up to two years
  Subjects underwent radical resection from the start until the date of the first documented tumor into recurrence or death from any cause, whichever occurred first
Overall survival (OS) | Up to two years
  Defined as the time from enrollment to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Zhongguo Zhou, Principal Investigator — Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou M, Wang H, Zeng X, Yin P, Zhu J, Chen W, Li X, Wang L, Wang L, Liu Y, Liu J, Zhang M, Qi J, Yu S, Afshin A, Gakidou E, Glenn S, Krish VS, Miller-Petrie MK, Mountjoy-Venning WC, Mullany EC, Redford SB, Liu H, Naghavi M, Hay SI, Wang L, Murray CJL, Liang X. Mortality, morbidity, and risk factors in China and its provinces, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2019 Sep 28;394(10204):1145-1158. doi: 10.1016/S0140-6736(19)30427-1. Epub 2019 Jun 24. PMID 31248666
- [Background] Siegel RL, Miller KD, Wagle NS, Jemal A. Cancer statistics, 2023. CA Cancer J Clin. 2023 Jan;73(1):17-48. doi: 10.3322/caac.21763. PMID 36633525
- [Background] Akateh C, Black SM, Conteh L, Miller ED, Noonan A, Elliott E, Pawlik TM, Tsung A, Cloyd JM. Neoadjuvant and adjuvant treatment strategies for hepatocellular carcinoma. World J Gastroenterol. 2019 Jul 28;25(28):3704-3721. doi: 10.3748/wjg.v25.i28.3704. PMID 31391767
- [Background] Zhang T, Zhang L, Xu Y, Lu X, Zhao H, Yang H, Sang X. Neoadjuvant therapy and immunotherapy strategies for hepatocellular carcinoma. Am J Cancer Res. 2020 Jun 1;10(6):1658-1667. eCollection 2020. PMID 32642282
- [Background] Papadopoulos KP, Harb W, Peer CJ, Hua Q, Xu S, Lu H, Lu N, He Y, Xu T, Dong R, Gong J, Liu D. First-in-Human Phase I Study of Envafolimab, a Novel Subcutaneous Single-Domain Anti-PD-L1 Antibody, in Patients with Advanced Solid Tumors. Oncologist. 2021 Sep;26(9):e1514-e1525. doi: 10.1002/onco.13817. Epub 2021 May 27. PMID 33973293
- [Background] Chen M, Jiang M, Wang X, Shen L, Li J. Envafolimab - first PD-1/PD-L1 antibody to be administered by subcutaneous injection for microsatellite instability-high or deficient mismatch repair advanced solid tumors. Expert Opin Biol Ther. 2022 Oct;22(10):1227-1232. doi: 10.1080/14712598.2022.2125799. Epub 2022 Sep 20. PMID 36124972
- [Background] Shimizu T, Nakajima TE, Yamamoto N, Yonemori K, Koyama T, Kondo S, Sunakawa Y, Izawa N, Horie Y, Xiang S, Xu S, Qin L, Gong J, Liu D. Phase I study of envafolimab (KN035), a novel subcutaneous single-domain anti-PD-L1 monoclonal antibody, in Japanese patients with advanced solid tumors. Invest New Drugs. 2022 Oct;40(5):1021-1031. doi: 10.1007/s10637-022-01287-7. Epub 2022 Aug 6. PMID 35932387
- [Background] Huang X, Xu L, Ma T, Yin X, Huang Z, Ran Y, Ni Y, Bi X, Che X. Lenvatinib Plus Immune Checkpoint Inhibitors Improve Survival in Advanced Hepatocellular Carcinoma: A Retrospective Study. Front Oncol. 2021 Nov 16;11:751159. doi: 10.3389/fonc.2021.751159. eCollection 2021. PMID 34868952